CLINICAL TRIAL: NCT00407095
Title: An Open Label SLV308 Safety Extension to Study S308.3.002 in Patients With Parkinson's Disease Experiencing Motor Fluctuations.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S308.3.007; 2006-005183-91 (EudraCT Number); 00407095 (Other Grant/Funding Number: NCT/NIH)
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Stage Parkinson's Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — pardoprunox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pardoprunox

INTERVENTIONS:
Drug: Pardoprunox — 12-42 mg/day

SUMMARY:
This study is a multicenter, 9 months, open label extension study for all patients who are willing and eligible to continue from the pivotal, double-blind S308.3.002 study.

ELIGIBILITY:
Inclusion Criteria Patients who have completed S308.3.002 trial Exclusion Criteria Patients with medically relevant abnormal findings (ECG, physical examination, Aes) at end of the maintenance phase (visit M6, week 24) of study S308.3.002

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety: laboratory data, adverse events, vital signs, ECG | 36 weeks

SECONDARY OUTCOMES:
On' and 'off' time recording, UPDRS parts 1-4, CGI-improvement, PDQ-39 total score: all change from baseline | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erik Vanleeuwen, Study Director — Abbott Products
Locations (87):
- United States (14):
  - S308.3.007 Site # 220, La Jolla, California
  - S308.3.007 Site # 211, San Francisco, California
  - S308.3.007 Site # 214, Fort Lauderdale, Florida
  - S308.3.007 Site # 218, Gainsville, Florida
  - S308.3.007 Site # 213, Tampa, Florida
  - S308.3.007 Site # 219, Augusta, Georgia
  - S308.3.007 Site # 221, Chicago, Illinois
  - S308.3.007 Site # 216, Kansas City, Kansas
  - S308.3.007 Site # 224, Lexington, Kentucky
  - S308.3.007 Site # 212, East Lansing, Michigan
  - S308.3.007 Site # 217, St Louis, Missouri
  - S308.3.007 Site # 222, Durham, North Carolina
  - S308.3.007 Site # 210, Tledo, Ohio
  - S308.3.007 Site # 215, Houston, Texas
- S308.3.007 Site # 223, Birmingham, Albania
- Argentina (10):
  - S308.3.007 Site # 100, Buenos Aires
  - S308.3.007 Site # 101, Buenos Aires
  - S308.3.007 Site # 102, Buenos Aires
  - S308.3.007 Site # 103, Buenos Aires
  - S308.3.007 Site # 106, Buenos Aires
  - S308.3.007 Site # 107, Buenos Aires
  - S308.3.007 Site # 109, Buenos Aires
  - S308.3.007 Site # 105, Córdoba
  - S308.3.007 Site # 104, Mar del Plata
  - S308.3.007 Site # 108, Santa Fe
- Brazil (11):
  - S308.3.007 Site # 114, Alto da Glória
  - S308.3.007 Site # 113, Belo Horizonte
  - S308.3.007 Site # 112, Campinas
  - S308.3.007 Site # 116, Marília
  - S308.3.007 Site # 111, Porto Alegre
  - S308.3.007 Site # 118, Porto Alegre
  - S308.3.007 Site # 117, Ribeirão Preto
  - S308.3.007 Site # 119, Salvador
  - S308.3.007 Site # 115, Sâo Paulo
  - S308.3.007 Site # 110, São Paulo
  - S308.3.007 Site # 125, São Paulo
- Bulgaria (5):
  - S308.3.007 Site # 123, Plovdiv
  - S308.3.007 Site # 120, Sofia
  - S308.3.007 Site # 121, Sofia
  - S308.3.007 Site # 122, Sofia
  - S308.3.007 Site # 124, Sofia
- Canada (10):
  - S308.3.007 Site # 136, Calgary
  - S308.3.007 Site # 137, Greenfield Park
  - S308.3.007 Site # 133, Halifax
  - S308.3.007 Site # 132, Markham
  - S308.3.007 Site # 130, Montreal
  - S308.3.007 Site # 134, Ottawa
  - S308.3.007 Site # 138, Peterborough
  - S308.3.007 Site # 135, Sainte-Anne
  - S308.3.007 Site # 139, Toronto
  - S308.3.007 Site # 131, Windsor
- Chile (4):
  - S308.3.007 Site # 140, Santiago
  - S308.3.007 Site # 141, Santiago
  - S308.3.007 Site # 143, Santiago
  - S308.3.007 Site # 142, Valdivia
- Colombia (5):
  - S308.3.007 Site # 151, Bogotá
  - S308.3.007 Site # 152, Bogotá
  - S308.3.007 Site # 153, Bogotá
  - S308.3.007 Site # 154, Bogotá
  - S308.3.007 Site # 150, Medellín
- S308.3.007 Site # 160, Riga, Latvia
- Lithuania (3):
  - S308.3.007 Site # 172, Kaunas
  - S308.3.007 Site # 170, Vilnius
  - S308.3.007 Site # 171, Vilnius
- Peru (5):
  - S308.3.007 Site # 184, Bellavista Callao
  - S308.3.007 Site # 180, Lima
  - S308.3.007 Site # 181, Lima
  - S308.3.007 Site # 182, Lima
  - S308.3.007 Site # 183, Lima
- Russia (9):
  - S308.3.007 Site # 193, Kazan'
  - S308.3.007 Site # 190, Moscow
  - S308.3.007 Site # 194, Moscow
  - S308.3.007 Site # 197, Moscow
  - S308.3.007 Site # 191, Saint Petersburg
  - S308.3.007 Site # 192, Saint Petersburg
  - S308.3.007 Site # 195, Saint Petersburg
  - S308.3.007 Site # 198, Saint Petersburg
  - S308.3.007 Site # 196, Yaroslavl
- Ukraine (9):
  - S308.3.007 Site # 204, Dnipro
  - S308.3.007 Site # 206, Kharkiv
  - S308.3.007 Site # 201, Kyiv
  - S308.3.007 Site # 202, Kyiv
  - S308.3.007 Site # 205, Lviv
  - S308.3.007 Site # 203, Poltava
  - S308.3.007 Site # 208, Simferopol
  - S308.3.007 Site # 200, Vinnytsia
  - S308.3.007 Site # 207, Zaporozhya